CLINICAL TRIAL: NCT02846207
Title: Study of Effects and Mechanisms of Yiqi Huoxue Demolition and Recipes on Recovery Stage of Cerebral Infarction
Brief Title: Yiqi Huoxue Demolition and Recipes on Recovery Stage of Cerebral Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Collaborators: Xingtai People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015CB554401
Record Dates: First submitted 2016-03-20; First posted 2016-07-27 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Cerebral Infarction
Keywords: cerebral infarction; syndrome of qi deficiency and blood stasis; Buyanghuanwu decoction; clinical effects and mechanisms
MeSH Terms: conditions — Cerebral Infarction | interventions — yiki-huoxue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Yiqi huoxue group (Experimental): Buyang Huanwu decoction , which includes: Astragalus 60g, Radix Paeoniae Rubra 15g, ligusticum wallichii 12g, angelica sinensis 20g, earthworm 12g, flos carthami 12g and peach seed 12g. Oral administration, twice one day, for 12weeks.
  Interventions: Drug: Yiqi huoxue
- Yiqi group (Experimental): Astragalus 60g. Oral administration, twice one day, for 12weeks.
  Interventions: Drug: Yiqi group
- Huoxue group (Experimental): Radix Paeoniae Rubra 15g, ligusticum wallichii 12g, angelica sinensis 20g, earthworm 12g, flos carthami 12g and peach seed 12g. Oral administration, twice one day, for 12weeks.
  Interventions: Drug: Huoxue group
- placebo group (Placebo Comparator): dextrin, Oral administration, twice one day, for 12weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Yiqi huoxue — Buyang Huanwu demolition, which includes: Astragalus 60g, Radix Paeoniae Rubra 15g, ligusticum wallichii 12g, angelica sinensis 20g, earthworm 12g, flos carthami 12g and peach seed 12g. Oral administration, twice one day, for 12weeks.
  Other Names: tonifying Qi and activating blood
  Arms: Yiqi huoxue group
Drug: Yiqi group — Astragalus 60g.Oral administration, twice one day, for 12weeks.
  Other Names: tonifying qi; benefiting qi
  Arms: Yiqi group
Drug: Huoxue group — Radix Paeoniae Rubra 15g, ligusticum wallichii 12g, angelica sinensis 20g, earthworm 12g, flos carthami 12g and peach seed 12g. Oral administration, twice one day, for 12weeks.
  Other Names: activating blood
  Arms: Huoxue group
Drug: placebo — Dextrin,oral administration, twice one day, for 12weeks.
  Other Names: a soothing restorative agency
  Arms: placebo group

SUMMARY:
This clinical research is based on the fundamentals of using Chinese medicine, which will improve Qi and promote blood circulation, to treat patients in the recuperating stages of cerebral infarction with deficiency in Qi and blood stasis syndrome. By assimilating Chinese medical theory, this research aims to study the biological basics of the stroke and the cause for the deficiency in Qi and blood stasis syndrome; explore the therapeutic mechanism of the treatment methods; as well as ascertaining the relationship between Qi, blood and blood vessels.

DETAILED DESCRIPTION:
Cerebral infarction, or ischemic stroke, is a common yet challenged illness with four telltale signs (high occurrence rate, high incapacitate rate, high mortality rate, and high recurrence rate), posing not only a threat to a man's health and life, but also imposing a burden to the society and his loved ones. As such, seeking a cure has always been the hot topic in this field of research. With regard to the illness' high incapacitate and recurrence rates, it has become apparent that the treatment methods used in the recuperating stages of stroke are very significant to the patient, allowing him the chance to regain his health and increase his quality of life. In Chinese medical terms, the pathogenesis key of stroke is a deficiency in the vitals of the body coupled with superficiality extremities. As such, in the recuperating stage of the stroke, a lack of Qi accompanied with blood stasis syndrome is often observed. Hence, improving Qi and promoting blood circulation is essential during treatment. Research further supports that this treatment method is highly effective in treating cerebral infarction, but the mechanism involved is still incomprehensible, largely due to the fact that the pathology of cerebral infraction is highly complicated, and that Chinese medicine is multi-leveled, multi-channeled, with multi-targets. To further study the relationship of Qi and blood in cerebral infraction, patients in the recuperating stages with deficiency in Qi and blood stasis underwent observation in a double blind clinical research. The patients were sorted in random into groups: improving Qi group, promoting blood circulation group, improving Qi and promoting blood circulation group, and the control group. Each group of patients was given the standard Western medicine treatment, coupled with Chinese medicine treatments with respect to their sorted groupings. The treatment lasts for 12 weeks and 360 clinical cases were studied. Testing methods used include enzyme linked immunosorbent assay, Western Blot, FQ RT-PCR, LC-MS, and radiology. Through the relations between Neurotransmitter - endocrine hormone - immune cytokine network, blood rheology, vascular structure and endothelial function, interactions involving vasoactive substances with vascular endothelium and blood cells, it is hoped that the biological basis of cerebral infraction's deficiency in Qi and blood stasis syndrome can be deciphered. This will aid in the understanding of the whole process of causing the syndrome, deciphering the therapeutic mechanism involved during treatment, as well as determining the relationship between Qi, blood and blood vessels.

ELIGIBILITY:
Inclusion Criteria:

1. In accordance to the Western medicine diagnostic criteria for atherosclerotic thrombotic cerebral infarction;
2. In accordance to the Chinese medicine diagnostic criteria for stroke, with deficiency in Qi and blood stasis syndrome;
3. In accordance to Stroke's diagnostic scale factor standards: asthenic Qi syndrome ≥ 10 points, blood stasis ≥ 10 points;
4. Within the recuperating stage of the illness (2 weeks to 6 months);
5. National Institutes of Health Stroke Scale (NIHSS) with a score of 3-22 points;
6. Ages within 35-80;
7. Signature of consent to participate in the research.

Exclusion Criteria:

1. Patients suffering from transient ischemic attack (TIA), subarachnoid haemorrhage and cerebral haemorrhage;
2. Patients suffering from cerebral embolism due to superficiality extremities caused by rheumatic heart disease, coronary heart disease and other heart diseases coupled with atrial fibrillation; stroke patients caused by brain tumor, head trauma, blood diseases, etc;
3. Pregnant women or women planning for pregnancy, women with positive urine pregnancy test, and lactating women;
4. Patients with severe hepatic and renal dysfunction, severe disease of the hematopoietic system, highly active ulcer and bleeding tendency, severe disease of the endocrine system, severe bone and joint disease, and arrhythmia patients with great clinical significance;
5. Patients with mental impairment, or mental disability, or severely deaf, or unconscious, or being uncooperative during inspection;
6. Patients with known allergies to the medicine used, as well as overly sensitive patients;
7. Patients that underwent clinical trials within the past 3 months.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
National Institute of Health Stroke Scale | 12 weeks
  NIHSS

SECONDARY OUTCOMES:
Modified Rankin scale | 12 weeks
  0-5scales
Barthel index | 12 weeks
  0-100scales

CONTACTS AND LOCATIONS:
Overall Officials: Liu Xiangzhe, PHD,MD, Principal Investigator — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine; Wang Jianhua, PHD,MD, Principal Investigator — Xingtai People's Hospital
Locations (3):
- China (3):
  - Dongfang Hospital, Beijing, Beijing Municipality
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Henan Univerisity of TCM, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li Y, Wang D, Guo R, Ma B, Miao L, Sun M, He L, Lin L, Pan Y, Ren J, Liu J. Neuroprotective effect of Astragali Radix on cerebral infarction based on proteomics. Front Pharmacol. 2023 Jun 9;14:1162134. doi: 10.3389/fphar.2023.1162134. eCollection 2023. PMID 37361203